CLINICAL TRIAL: NCT03122119
Title: Effectiveness of Ultrasound Guided Platelet Rich Plasma Injections in the Sacroiliac Joint to Relieve Low Back Pain
Brief Title: Effectiveness of Ultrasound Guided Platelet Rich Plasma Injections in the Sacroiliac Joint
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Star Spine and Sport (Other)
Responsible Party: Principal Investigator, Douglas Hemler, Principal Investigator, Star Spine and Sport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP SIJ Injection Ultrasound
Record Dates: First submitted 2017-04-16; First posted 2017-04-20 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Chronic Low Back Pain; Sacroiliitis; Sacroiliac; Backache; Platelet Rich Plasma; Platelet; Injection Site; Ultrasound Therapy; Complications; Treatment
Keywords: Sacroiliac; Joint Injection; Platelet Rich Plasma; Ultrasound; Low Back Pain
MeSH Terms: conditions — Sacroiliitis; Back Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Platelet Rich Plasma Joint Injection (Experimental): Venous blood will be drawn from the patient receiving injection treatment. It will be spun down to form PRP and reinjected back into the SI joint.
  Interventions: Drug: Platelet Rich Plasma Joint Injection

INTERVENTIONS:
Drug: Platelet Rich Plasma Joint Injection — 30 to 50 milliliters of venous blood will be drawn from the patients arm with a 19 gauge ¾ inch needle using universal precautions. The venous blood will be mixed with 8 milliliters of anticoagulant citrate dextrose solution-A (ACD-A). The anti-coagulated blood will then be centrifuged for 15 minutes at 3200 revolutions per minute in the office centrifuge. This will allow plasma to separate from blood cells. The portion of centrifuged blood deficient in platelets will be extracted and discarded. Once the needle is visualized entering the joint capsule via ultrasound guidance and the physician feels resistance provided by the capsule and ligaments, 3 milliliters of PRP extract will be injected (3 inch, 22 gauge needle) into the sacroiliac joint. The needles will be properly disposed.
  Other Names: PRP Joint Injection; PRP

SUMMARY:
This prospective study will be quantitatively analyzing the effectiveness of platelet-rich-plasma (PRP) injections into the sacroiliac (SI) joint in relieving sacroiliitis and low back pain originating from the SI joint. The effectiveness of PRP injections on joint pain has been well studied in the knee and shoulder. PRP injections are performed on the SI joint commonly, but there is little research documenting their effectiveness when compared to other interventions. This study will be a small pilot study to aid in closing this knowledge gap. Additionally, these injections will be performed under ultrasound guidance. Ultrasound has been proven to be of equal reliability to fluoroscopy and has the advantage of shorter time to administer and no radiation. There will be one arm to this study. The data collected will be compared to existing studies on corticosteroid SI joint injection. The experimental arm consists of the PRP injection. The PRP will be injected into the joint using the exact same technique via physical exam, special tests, and ultrasound guidance as performed in our previous studies. The outcomes will be measured with the Numeric Rating Scale for Pain (NRS) and the Oswestry Disability Index (ODI) prior to the injection, immediately post-injection, 2 weeks, 4 weeks, 3 months, and 6 months post-injection. The investigators hypothesis is, "Platelet-Rich Plasma Injections in the Sacroiliac Joint using ultrasonography in conjunction with physical examination and Point of Maximal Tenderness will produce statistically significant pain relief for more than 3 months as measured by the Numeric Rating Scale for Pain (NRS) and Oswestry Disability Index (ODI)."

DETAILED DESCRIPTION:
PRP is not just an additional tool for physicians to use, but a potential treatment for underlying joint pathology. PRP is one of the closest treatments that exists for a definitive solution for inflammatory and degenerative joint disease. PRP is currently being used for dysfunction of the shoulder joint, knee joint, sacroiliac joint, facet joints, intervertebral discs, rotator cuff, hamstrings, and others. It has been extensively researched for osteoarthritis, tendon, and ligament injury of the knee, but little research has documented the short or long-term effects on the sacroiliac joint. A brief search on PubMed provides only two articles, one of which is a case study, and neither were performed in the United States. PRP is the future of orthopedics and physical medicine as well as a gateway to curing degenerative and inflammatory joint disease.

Furthermore, the use of ultrasound guided injections has helped increase the success rate because it provides a method for visualizing the path of the needle to a precise location. In recent studies, authors have indicated the use of a curvilinear transducer to be the most successful, as well as injections administered to the lower one third of the sacroiliac joint, to be adequately effective in diagnosing and treating sacroiliac joint pain. Disadvantages surrounding fluoroscopy include inconvenience, cost, radiation, and exposure to contrast media. Arranging the procedure can take extensive time and resources. The procedure can be costly for the patient, especially if it does not produce long-term results, and radiation exposure can have long-term consequences for the patient's health, rendering it a questionable treatment for chronic low back pain. As ultrasound guided and fluoroscopic sacroiliac joint injections present themselves as front-runners for diagnosis and treatment of sacroiliac joint-induced low back pain, the benefits and downsides to both are heavily weighed and compared. The next step moving forward in the treatment of the SI joint is administering PRP injections while utilizing ultrasonography for image guidance. The investigators believe this combination will provide the most immediate and long term benefit to patients as well as fewer risks from medications, corticosteroids, and fewer risks and downsides from fluoroscopy, such as radiation and cost.

Experimental design will be a nonrandomized trial (or quasi-experiment). The specific study design to be used is pretest-posttest design. The independent variable will be the PRP injection. The dependent variables of interest include the NRS and Oswestry Disability Index (ODI) recording pre-injection, immediately post-injection, 2 weeks, 4 weeks, 3 months, 6 months post-injection.

Most studies in the past look at short-term and moderate-term results up to approximately six months to one year. Many studies state a limitation to their data is the lack of long-term investigation into pain, disability, and function more than 12 months. This is partly due to losing patients to follow up. Patients whose pain resolved have no reason to return for further evaluation.

The investigators will take measures to avoid study bias and confounding by ensuring patients have been correctly diagnosed with sacroiliitis via special tests and physical examination as well as PMT. Additionally, to avoid confounding, the investigators will not administer PRP injections to patients who have had a corticosteroid injection in the SI joint within the last three months or received significant benefit from a corticosteroid injection. The efficacy of corticosteroids in the joint begin to dwindle starting at approximately three months.

This information will be recorded in each patient's chart as well as an Excel file only accessible to key personnel working on the study. The following data will be recorded form each patient: current pain scale using the NRS and their functionality using the ODI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sacroiliitis
* Age 18 to 80 years old
* Chronic low back pain
* SI joint pathology is the predominant source of pain
* Positive Fortin Finger Test (PMT)
* Joint anatomy is identifiable using ultrasonography
* Patient has no other comorbidities that contraindicate the procedure
* Patient has attempted physical therapy and corticosteroid injections with local anesthetic -Previous injections of lidocaine and corticosteroid provided at least minor immediate relief
* Patient must not have had a corticosteroid injection in the SI joint within the last three months
* Patient must consent to the procedure

Exclusion Criteria:

* Patients under the age of 18 (Subjects under the age of 18 will not be included in this study due to the continued growth and development of their joints and unstudied effects on children.)
* Over the age of 80
* Multiple pain sources and multifactorial pain sources that complicated or confound diagnosing the SI joint as the primary and predominant pain generator that may contribute to low back pain (including but not limited to: lumbar diagnosis, lumbar radiculopathy, intra or extra-articular hip pathology to include acetabulum and femoral head, lumbo-sacral joint pathology, intervertebral disk disease, spondylolisthesis/spondylosis/spondylolysis of lumbar vertebra)
* Immunosuppressed/immune compromised
* Underlying comorbidities that contraindicate the procedure (including but not limited to polycythemia, coagulation disorder, or malignancy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hemler, MD, Principal Investigator — Star Spine and Sport, Rocky Vista University College of Osteopathic Medicine
Locations (1):
- Star Spine and Sport, Golden, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarzer AC, Aprill CN, Bogduk N. The sacroiliac joint in chronic low back pain. Spine (Phila Pa 1976). 1995 Jan 1;20(1):31-7. doi: 10.1097/00007632-199501000-00007. PMID 7709277
- [Background] Dreyfuss P, Dreyer SJ, Cole A, Mayo K. Sacroiliac joint pain. J Am Acad Orthop Surg. 2004 Jul-Aug;12(4):255-65. doi: 10.5435/00124635-200407000-00006. PMID 15473677
- [Background] Vleeming A, Schuenke MD, Masi AT, Carreiro JE, Danneels L, Willard FH. The sacroiliac joint: an overview of its anatomy, function and potential clinical implications. J Anat. 2012 Dec;221(6):537-67. doi: 10.1111/j.1469-7580.2012.01564.x. Epub 2012 Sep 19. PMID 22994881
- [Background] Lennard T, Fortin J. Sacroiliac Joint Injection and Arthrographic Imaging Correlation In: Physiatric Procedures in Clinical Practice. Philadelphia: Hanley & Belfus, 1995. 242-253.
- [Background] Harmon D, O'Sullivan M. Ultrasound-guided sacroiliac joint injection technique. Pain Physician. 2008 Jul-Aug;11(4):543-7. PMID 18690282
- [Background] Singla V, Batra YK, Bharti N, Goni VG, Marwaha N. Steroid vs. Platelet-Rich Plasma in Ultrasound-Guided Sacroiliac Joint Injection for Chronic Low Back Pain. Pain Pract. 2017 Jul;17(6):782-791. doi: 10.1111/papr.12526. Epub 2016 Dec 1. PMID 27677100
- [Background] Sakata R, Reddi AH. Platelet-Rich Plasma Modulates Actions on Articular Cartilage Lubrication and Regeneration. Tissue Eng Part B Rev. 2016 Oct;22(5):408-419. doi: 10.1089/ten.TEB.2015.0534. Epub 2016 Jun 27. PMID 27109909
- [Background] Ko GD, Mindra S, Lawson GE, Whitmore S, Arseneau L. Case series of ultrasound-guided platelet-rich plasma injections for sacroiliac joint dysfunction. J Back Musculoskelet Rehabil. 2017;30(2):363-370. doi: 10.3233/BMR-160734. PMID 27392848
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Zanon G, Combi F, Combi A, Perticarini L, Sammarchi L, Benazzo F. Platelet-rich plasma in the treatment of acute hamstring injuries in professional football players. Joints. 2016 Jun 13;4(1):17-23. doi: 10.11138/jts/2016.4.1.017. eCollection 2016 Jan-Mar. PMID 27386443
- [Background] Andia I, Rubio-Azpeitia E, Maffulli N. Platelet-rich plasma modulates the secretion of inflammatory/angiogenic proteins by inflamed tenocytes. Clin Orthop Relat Res. 2015 May;473(5):1624-34. doi: 10.1007/s11999-015-4179-z. PMID 25670657
- [Background] Chen CP, Lew HL, Tsai WC, Hung YT, Hsu CC. Ultrasound-guided injection techniques for the low back and hip joint. Am J Phys Med Rehabil. 2011 Oct;90(10):860-7. doi: 10.1097/PHM.0b013e318228c084. PMID 21844793
- [Background] Chang WH, Lew HL, Chen CP. Ultrasound-guided sacroiliac joint injection technique. Am J Phys Med Rehabil. 2013 Mar;92(3):278-9. doi: 10.1097/PHM.0b013e318278d108. No abstract available. PMID 23221672
- [Background] Hassan AS, El-Shafey AM, Ahmed HS, Hamed MS. Effectiveness of the intra-articular injection of platelet rich plasma in the treatment of patients with primary knee osteoarthritis. The Egyptian Rheumatologist. 2015;37(3):119-124.
- [Background] Kirchner F, Anitua E. Intradiscal and intra-articular facet infiltrations with plasma rich in growth factors reduce pain in patients with chronic low back pain. J Craniovertebr Junction Spine. 2016 Oct-Dec;7(4):250-256. doi: 10.4103/0974-8237.193260. PMID 27891035
- [Background] Raeissadat SA, Rayegani SM, Hassanabadi H, Fathi M, Ghorbani E, Babaee M, Azma K. Knee Osteoarthritis Injection Choices: Platelet- Rich Plasma (PRP) Versus Hyaluronic Acid (A one-year randomized clinical trial). Clin Med Insights Arthritis Musculoskelet Disord. 2015 Jan 7;8:1-8. doi: 10.4137/CMAMD.S17894. eCollection 2015. PMID 25624776
- [Background] Gobbi A, Karnatzikos G, Mahajan V, Malchira S. Platelet-rich plasma treatment in symptomatic patients with knee osteoarthritis: preliminary results in a group of active patients. Sports Health. 2012 Mar;4(2):162-72. doi: 10.1177/1941738111431801. PMID 23016084
- [Background] Vianin M. Psychometric properties and clinical usefulness of the Oswestry Disability Index. J Chiropr Med. 2008 Dec;7(4):161-3. doi: 10.1016/j.jcm.2008.07.001. PMID 19646379
- [Background] Joshi VD, Raiturker PP, Kulkarni AA. Validity and reliability of English and Marathi Oswestry Disability Index (version 2.1a) in Indian population. Spine (Phila Pa 1976). 2013 May 15;38(11):E662-8. doi: 10.1097/BRS.0b013e31828a34c3. PMID 23380824
- [Background] Copay AG, Cher DJ. Is the Oswestry Disability Index a valid measure of response to sacroiliac joint treatment? Qual Life Res. 2016 Feb;25(2):283-292. doi: 10.1007/s11136-015-1095-3. Epub 2015 Aug 6. PMID 26245709
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Barile A, La Marra A, Arrigoni F, Mariani S, Zugaro L, Splendiani A, Di Cesare E, Reginelli A, Zappia M, Brunese L, Duka E, Carrafiello G, Masciocchi C. Anaesthetics, steroids and platelet-rich plasma (PRP) in ultrasound-guided musculoskeletal procedures. Br J Radiol. 2016 Sep;89(1065):20150355. doi: 10.1259/bjr.20150355. Epub 2016 Jul 7. PMID 27302491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 participants between the ages of 18 and 80 years old with chronic low back pain and a diagnosis of sacroiliitis were selected for this single center clinical trial. The Setting was a privately owned physical medicine and rehabilitation clinic.
Period: Overall Study
Arm/Group | Platelet Rich Plasma Joint Injection
Started | 51
Completed | 50
Not Completed | 1
Not completed — Did not meet eligibility critria | 1

BASELINE CHARACTERISTICS:
Population: not different from the assignment in participant flow
Arm/Group | Platelet Rich Plasma Joint Injection
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline Pain - Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Numeric Rating Scale for pain measures pain levels on a scale of 0 to 10 with 0 being no pain and 10 being the worst pain possible.
  units on a scale | 6.05 (1.69)
Baseline - Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: units on a scale] — Oswestry Disability Index measures amount of disability with a range from 0 to 50 with 0 being no disability and 50 being completely disabled.
  units on a scale | 37.86 (14.65)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale for Pain (NRS)
Description: Defined as a numeric scale for pain from 0 to 10. 0 demonstrates no pain and 10 demonstrates severe pain or significant impact on activities of daily living.
Time Frame: Change from baseline compared to 6 months post injection
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Platelet Rich Plasma Joint Injection
Number analyzed (Participants) | 50
units on a scale
  Baseline pain to 2-week post injection pain | 1.08 [0.45 to 1.72]
  Baseline pain to 4-week post injection pain | 1.58 [1.02 to 2.14]
  Baseline pain to 3-month post injection pain | 1.69 [1.02 to 2.37]
  Baseline pain to 6-month post injection pain | 1.94 [1.14 to 2.78]

2. Primary Outcome: Oswestry Disability Index (ODI)
Description: Standardized questionnaire which asks 10 questions to assess impact on activities of daily living. Minimum score is 0, maximum score is 50. Higher scores mean worse outcome or more impact on function.
Time Frame: Change from baseline compared to 6 months post injection
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Platelet Rich Plasma Joint Injection
Number analyzed (Participants) | 50
units on a scale
  Baseline disability to 2-week post-injection disability | 4.72 [2.27 to 7.17]
  Baseline disability to 4-week post-injection disability | 7.14 [4.49 to 9.78]
  Baseline disability to 3-month post-injection disability | 8.78 [4.62 to 12.93]
  Baseline disability to 6-month post-injection disability | 9.79 [6.06 to 13.52]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Platelet Rich Plasma Joint Injection
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT03122119/Prot_SAP_002.pdf